CLINICAL TRIAL: NCT07202780
Title: Examination of the Relationship Between Mechanical Properties of Respiratory and Lower Extremity Muscles, Respiratory Function, Fatigue, and Anxiety-Depression in Patients With Multiple Sclerosis
Brief Title: The Relationship Between Mechanical Properties of Respiratory and Lower Extremity Muscles and Other Parameters in Multiple Sclerosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Burcu Bağcı, Assisant Prof., Sanko University
Other Study IDs: Burcu3
Record Dates: First submitted 2025-09-16; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis; Breath Tests; MyotonPRO
Keywords: multiple skleroz; breath test; myoton pro
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multiple sclerosis people: Individuals diagnosed with MS were included
- healthy individuals: healthy individuals were included

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease characterised by deterioration in the mechanics of the lower extremities and respiratory muscles and a decrease in respiratory function. Fatigue and depression are among the most common symptoms. The aim of this study is to investigate the potential effect of the mechanical properties of the lower extremity and respiratory muscles on respiratory function, fatigue, and anxiety-depression. The sample will consist of 29 MS patients who meet the inclusion and exclusion criteria and volunteer to participate in the study. The sociodemographic data of the individuals will be recorded. Subsequently, the Pulmonary Dysfunction Index (PDI), Modified Medical Research Council Scale (mMRC), Expanded Disability Status Scale (EDSS), Fatigue Severity Scale (FSS), and Hospital Anxiety and Depression Scale (HADS) will be administered to the individuals. The mechanical properties of the accessory respiratory and lower extremity muscles will be recorded using a digital palpation device, and respiratory function and respiratory muscle strength values will be recorded using a portable spirometer. Lower extremity function and strength will be assessed using the 30-second sit-to-stand test. At the end of the study, the level of association between the mechanical properties of the auxiliary respiratory and lower extremity muscles and respiratory function, respiratory muscle strength, fatigue, and depression will be evaluated. The SPSS software package will be used for data analysis. A significance level of p˂0.05 will be accepted. Furthermore, this study will determine the relationship between the mechanical properties of respiratory and lower extremity muscles in MS and provide a different perspective on the clinical management of the disease.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory disease characterised by demyelination and axonal degeneration in the central nervous system, leading to various motor and sensory impairments. Symptoms are classified as cognitive, sensory, and motor, with the most common symptoms including loss of muscle control, muscle weakness, abnormal muscle tone, ataxia, depression, and fatigue. These impairments frequently affect balance and gait, leading to the disabling consequences of the disease. The muscle groups most affected in individuals with MS are the lower extremities, which exhibit significant reductions in muscle strength and function. Research shows that in the early stages of MS, muscle strength in the lower extremities can decrease by approximately 25% compared to healthy controls, with marked deficiencies in muscle activation and increased fatigue. Studies have shown that quadriceps strength is significantly reduced, which can lead to difficulties in walking and maintaining balance. Furthermore, in MS patients, the coactivation patterns of lower limb muscles during walking change, indicating a compensatory mechanism in response to decreased muscle strength. This coactivation can lead to inefficient movement patterns, further exacerbating fatigue and functional limitations.

Fatigue is another important symptom associated with MS and affects both voluntary and involuntary muscle contractions. Approximately 65% of individuals with MS report fatigue, and 40% describe fatigue as the most disabling symptom. However, despite the prevalence of fatigue in MS, its exact mechanisms remain unclear. It has been suggested that there may be a correlation between fatigue and increased central arousal to compensate for reduced central activation, and depression has also been reported as a factor that increases fatigue. Fatigue is not only a result of muscle weakness but also involves central mechanisms that impair motor control and muscle activation.

Disability in MS is associated with reduced mobility, abnormal gait mechanics, impaired balance and muscle weakness, as well as cognitive and autonomic dysfunction. These impairments typically reduce functional capacity, increase fatigue, reduce independence in activities of daily living, and consequently increase the risk of secondary diseases such as coronary heart disease, diabetes, and obesity. Therefore, a good understanding of fatigue and the mechanical properties of muscle in these patients may play an important role in disease progression.

MS can affect the trunk and respiratory muscles as well as the lower extremities. Factors affecting respiratory function include muscle weakness, changes in muscle tone, motor coordination disorders, and postural abnormalities. In addition, MS can affect the centres responsible for respiratory function, leading to clinically significant changes in respiratory control. It has been reported that respiratory muscle weakness can be observed even in the early stages of MS. These studies highlight the complex effect of MS on respiratory function and respiratory muscle weakness.

In summary, MS is a multi-faceted disease that can affect the muscles of the lower extremities, particularly the quadriceps, as well as the trunk and respiratory muscles. These impairments can lead to significant functional limitations, affecting the mobility and overall quality of life of individuals with MS and potentially worsening the progression of the disease. Therefore, it is important to understand this condition well and take it into account in clinical management. However, lower limb and respiratory muscle mechanics, respiratory function, fatigue, and depression levels in individuals with MS have not been comprehensively investigated. Therefore, the aim of this study is to investigate the potential relationship between lower limb and respiratory muscle mechanics, respiratory function, fatigue, and anxiety-depression in individuals with MS.

Research Hypotheses:

H0: The mechanical properties of the respiratory and lower extremity muscles in individuals with multiple sclerosis have no effect on respiratory function, fatigue, and depression levels.

H1: The mechanical properties of the respiratory and lower extremity muscles in individuals with multiple sclerosis have an effect on respiratory function, fatigue, and depression levels.

This study will be conducted jointly by the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, SANKO University, and the Department of Neurology, Faculty of Medicine, SANKO University. MS patients who apply to the Neurology Outpatient Clinic of SANKO University Hospital and meet the inclusion criteria will be included in the study. Patients included in the study will be evaluated at the SANKO University Department of Physiotherapy and Rehabilitation Research Laboratory.

The study data were collected using the Case Report Form (CRF), Pulmonary Dysfunction Index (PDI), Modified Medical Research Council Scale (mMRC), Expanded Disability Status Scale (EDSS), Fatigue Severity Scale (FSS), and Hospital Anxiety and Depression Scale (HADS). Data contained in the Data Collection Form (DCF) will be obtained using the 30-second sit-to-stand functional assessment test (30sSTT) and laboratory measurement devices including the MyotonPro® digital palpation device (Myoton AS, Estonia) and a portable spirometer (Cosmed, Pony Fx, Rome, Italy).

The study data were collected using the Case Report Form (CRF), Pulmonary Dysfunction Index (PDI), Modified Medical Research Council Scale (mMRC), Expanded Disability Status Scale (EDSS), Fatigue Severity Scale (FSS), and Hospital Anxiety and Depression Scale (HADS). Data contained in the Data Collection Form (DCF) will be obtained using the 30-second sit-to-stand functional assessment test (30sSTT) and laboratory measurement devices including the MyotonPro® digital palpation device (Myoton AS, Estonia) and a portable spirometer (Cosmed, Pony Fx, Rome, Italy).

Healthy individuals of the same age group will be included in the study. The results of healthy individuals will be compared with the results of MS patients.

ELIGIBILITY:
Inclusion Criteria

* Having been diagnosed with MS according to the revised McDonald criteria followed at the Neurology Outpatient Clinic of Sanko University Hospital,
* Being between 18 and 50 years of age,
* Not having had an attack in the last 6 months,
* Having an EDSS score of 4.5 or below,
* To have given consent for the study.

Exclusion Criteria:

History of lower extremity surgery within the last 12 months,

* To have undergone physiotherapy within the last 6 months,
* Presence of current trauma or fracture involving the lower extremities,
* Presence of another neuro-musculoskeletal or pulmonary disease besides MS,
* Inability to cooperate with measurements and demonstrate compliance,
* Having received pulse steroid therapy or botulinum toxin/phenol injection within the last 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Having been diagnosed with MS according to the revised McDonald criteria followed at the Neurology Outpatient Clinic of Sanko University Hospital
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Neurological Disability Level: | 1 year
  The neurological disability level of individuals with MS will be determined using the Expanded Disability Status Scale (EDSS), a widely used scale. Developed by Kurke, it has been the most commonly used method for measuring disability in the field of MS for many years. The EDSS is used to measure the level of disability in MS. The validity and reliability of the EDSS in Turkish, particularly when used in conjunction with other scales to comprehensively assess disability in the context of MS, has been demonstrated in various studies. The EDSS is a 20-stage disease severity scale ranging from 0 (normal) to 10 (death due to MS).
Fatigue Severity Scale | 1 year
  The Fatigue Severity Scale (FSS) was first developed by Krupp et al. (1989). This scale was specifically designed to assess the severity of fatigue in patients with MS and other chronic conditions. Its validity and reliability in Turkish-speaking MS patients were demonstrated by Armutlu et al. (2007). The FSS consists of nine items that assess the impact of fatigue on daily functioning and overall quality of life, with responses measured on a seven-point Likert scale. In the self-administered version of the scale, each item is scored from 1 to 7 (1 = strongly disagree, 7 = strongly agree), and the total score is calculated as the average of the nine items. The lower the total score, the less fatigue is present. A commonly used cut-off value in clinical practice is a total score of 36 or higher, indicating significant fatigue.
The Hospital Anxiety and Depression Scale | 1 year
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess depression. Developed by Zigmond et al. (1983), this scale consists of 14 questions, seven measuring anxiety and seven measuring depression. A four-point Likert-type scale is used to answer each question. Each item is scored between 0 and 3, and the total score is calculated as the average of the seven items. The scale has been adapted into Turkish, and as a result of the validity and reliability study, the cut-off score for the anxiety subscale was found to be 10/11, and the cut-off score for the depression subscale was found to be 7/8. In our study, each HADS score for anxiety and depression will be considered as follows: 0-7 = normal, 8-10 = borderline abnormal, 11-21 = abnormal.
myoton pro | 1 year
  The muscles of the patients' lower extremities, including the Rectus Femoris, Vastus Lateralis, Vastus Medialis, Biceps Femoris, Semitendinosus, Gastrocnemius Medialis, and Gastrocnemius Lateralis, as well as the auxiliary respiratory muscles, including the Sternocleidomastoideus, M. Upper Trapezius, M. Pectoralis Major, M. Serratus Anterior, M. Rectus Abdominis, and M. External Oblique Abdominis will be assessed using the MyotonPro® (Myoton AS, Estonia) digital palpation device.
Assessment of Lower Limb Functionality and Muscle Strength | 1 years
  The 30-second sit-to-stand test (30s-OKT) will be used to measure lower limb functionality and muscle strength. The test, developed by Jones et al. (1999), is a functional assessment test. The 30sOKT has been validated as an effective measure of lower extremity strength, particularly in patients with MS, and has shown strong correlations with other functional assessments such as the Timed Up and Go (TUG) test and the 5-repetition sit-to-stand test (5STS). In our country, Özkeskin et al. (2023) applied this test to patients with MS and reported that the test-retest reliability was excellent (ICC > 0.80) and the concurrent validity (r > 0.05) was strong. Prior to the test, patients will rest for 30 minutes, and the physiotherapist administering the test will demonstrate how the test is performed to the patient. Patients will be seated upright on an armless chair (approximately 43 cm high) with their back against the wall, their
Assessment of Respiratory Muscle Strength: | 1 year
  In clinical practice, respiratory muscle strength is assessed based on the principle of measuring the pressure difference between inspiration and expiration. Maximal voluntary inspiratory (PImax) and expiratory (PEmax) pressures (MIP and MEP) are the most commonly used non-invasive methods for measuring respiratory muscle strength (ATS/ERS, 2022). Black and Hyatt (1969) stated that this technique can be used for health checks in patients and athletes of all ages. Pressure is measured by performing maximal inspiration (Müller manoeuvre) and expiration (Valsalva manoeuvre) through the mouth. The manoeuvre is typically performed at residual volume (RV) for MIP and total lung capacity (TLC) for MEP (Cotes et al., 2006; Ruppel, 2009). In our study, patients' intraoral pressure measurements will be taken using a Cosmed Pony FX model device (Italy).
  Measurements were performed in a sitting position with a nose clip. The Valsalva and Müller manoeuvr
A Spirometry Test (SFT) | 1 years
  involves the measurement of dynamic lung volumes and capacities over time during forced inspiration and expiration (Bartu-Saryal and Ulubay, 2012). In our study, SFT measurements will be performed using a Cosmed Pony FX model (Italy) portable spirometer.
  Patients will be informed about the PFT in advance, in accordance with measurement standards. To enable comparison with standard values, patients' gender, age, height, weight, and ethnicity (e.g., Caucasian) will be entered into the device. Tests will be performed in a seated position. At least 3 tests will be performed on each patient, and measurements will not be continued for cases that fail to perform the manoeuvre successfully after 8 tests. During the test, subjects will be asked to take 3-4 normal breaths and then take a deep inspiration, followed by a rapid and forceful expiration to expel all air (ATS/ERS, 2005). After three successful tests, the test with the highest sum of FVC and FEV1, as recommend

CONTACTS AND LOCATIONS:
Locations (1):
- Sanko University, Gaziantep, şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No